CLINICAL TRIAL: NCT07315711
Title: The Effect of Vascular Imaging Devices on the Success Rate of Peripheral Vascular Access in Pediatric Patients Undergoing Day-Case and Non-Operating Room Anesthesia Procedures
Brief Title: The Effect of Vascular Imaging Devices on Success Rates of Peripheral Vascular Access in Pediatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sibel Seçkin Pehlivan (Other)
Responsible Party: Sponsor-Investigator, Sibel Seçkin Pehlivan, Assistant Professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 2025/454
Record Dates: First submitted 2025-12-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Vascular Access in Pediatric Patients; Peptic Ulcer; Cataract; Crohn's Disease
Keywords: non-operating room anesthesia (NORA), peripheral vascular access, pediatric patienent
MeSH Terms: conditions — Peptic Ulcer; Cataract; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Pediatric patients undergoing peripheral vascular access with the use of a vascular imaging device. The intervention involves the application of real-time imaging guidance (e.g., near-infrared light or ultrasound) to facilitate successful and efficient cannulation.
- Control Group: Pediatric patients undergoing peripheral vascular access without the use of a vascular imaging device, relying on standard visual and palpation techniques.

SUMMARY:
The study was designed as a prospective, observational study. Pediatric patients under 18 years of age scheduled for peripheral vascular access placement during day-case surgery or non-operating room anesthesia (NORA) will be included. The primary outcomes include time to successful vascular access, number of attempts, and number of interventions (defined as each new skin entry of the needle). These outcomes will be compared between two groups: those who receive vascular access with the aid of a vascular imaging device and those in whom such a device is not used.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0-18 years scheduled for day-case surgery or non-operating room anesthesia (NORA)

Patients requiring peripheral vascular access (those with a need for intravenous access)

Patients whose parent or legal guardian can provide written informed consent

Patients suitable for vascular access using a vascular imaging device

Exclusion Criteria:

Patients requiring emergency surgery or urgent intervention

Patients whose parent or legal guardian cannot provide informed consent

Patients with local extremity problems such as infection, edema, or wound that prevent peripheral vascular access placement

-

Ages: 0 Days to 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 0-18 years scheduled for day-case surgery or non-operating room anesthesia (NORA)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The time to establish peripheral vascular access | pre-intervention/procedure/surgery
  The primary outcome measure is the time required to successfully establish peripheral vascular access, defined as the interval from the first needle insertion attempt to the confirmation of intravenous placement (e.g., blood return and/or free flow of saline). This metric will be recorded in seconds and compared between patients who receive vascular imaging assistance and those who do not.
number of attempts | pre-intervention/procedure/surgery
  The number of attempts refers to the total number of needle insertions required to achieve successful peripheral vascular access, with each attempt defined as a distinct skin puncture. An attempt is counted even if cannulation is not achieved. This outcome will be documented for each patient and compared between the group using vascular imaging devices and the group without such assistance.

SECONDARY OUTCOMES:
number of interventions (each new skin entry of the needle) | pre-intervention/procedure/surgery
  The number of interventions refers to the total count of new skin entries made with the needle during peripheral vascular access attempts. Each distinct insertion of the needle through the skin, regardless of whether it occurs during the same cannulation effort or a subsequent repositioning, is recorded as a separate intervention. This metric will be used to assess procedural invasiveness and will be compared between patients who undergo vascular access with versus without vascular imaging device assistance

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Seckin Pehlivan, Principal Investigator — Department of Anaesthesiology and Reanimation, Erciyes University, Kayseri, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University Hospital, Kayseri, Kayseri̇
  - Erciyes University Hospital, Kayseri

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and ethical considerations regarding patient confidentiality. Data are stored securely in accordance with local regulations, and dissemination is limited to aggregated results to protect the privacy of pediatric patients involved in the study.